CLINICAL TRIAL: NCT05900089
Title: Efficacy and Safety of SHR0302 in Patients With Relapsed/Refractory Peripheral T/NK Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCL-IIT-SHR0302
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — ivarmacitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR0302 Group A (Experimental)
  Interventions: Drug: SHR0302
- SHR0302 Group B (Experimental)
  Interventions: Drug: SHR0302
- SHR0302 Group C (Experimental)
  Interventions: Drug: SHR0302

INTERVENTIONS:
Drug: SHR0302 — SHR0302 will be administered orally as tablet. SHR0302 treatment will be continued until disease progression or intolerant adverse reactions

SUMMARY:
This is a non-randomized, open-label, Phase 1b clinical study to evaluate the safety, tolerability and anti-tumor efficacy of SHR0302 as monotherapy in patients with relapsed/refractory peripheral T/NK cell lymphoma. Around 7-18 patients will be subsequently enrolled into 3 different dose ascending cohorts. Additional 12-18 patients may be enrolled to further explore a selected dose defined by dose escalation cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18;
2. Pathologically confirmed T or NK cell lymphoma at the enrolling institution;
3. Measurable disease;
4. Relapse or refractory disease after at least 1 systemic therapy;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2 ；
6. With a life expectancy of ≥12 weeks;
7. Adequate bone marrow reserve and organ system functions;
8. Women of Childbearing Potential (WOBCP) must undergo a serum pregnancy test within seven days before the first medication and the results are negative. WOBCP or men and their WOBCP partners should agree to take effective contraceptive measures from the signing of ICF until 180 days after the last dose of the study drug is used;
9. Willing to provide written informed consent.

Exclusion Criteria:

1. Patient has undergone an allogeneic stem cell transplant. Or patient had autologous stem cell transplant within 6 months;
2. Any unsolved toxicity > Common Terminology Criteria for Adverse Events (CTCAE) grade 1 from previous anti-cancer therapy (except alopecia);
3. Central nervous system (CNS) or leptomeningeal lymphoma;
4. received any antitumor therapy within 28 days prior to the first drug use, or the first dose was given within five half-lives of the previous antitumor drug, whichever is shorter;
5. Major surgical procedures were performed within 28 days before the first dose of study treatment, or surgery was planned during the study period;
6. Diagnosed with any other malignancies ≤5 years prior to the first dose, early tumors cured after radical treatment were evaluated by PI and considered for exclusion or not;
7. History of psychotropic substance abuse or drug use;
8. Previous history of allergy to the investigational drug or its excipients;
9. Severe cardiovascular disease;
10. Significant impairment of lung function;
11. Active infections;
12. Pregnant or lactation;
13. Known GI disease or GI procedure that could interfere with the oral absorption of oral medications, including not well controlled refractory nausea, vomiting, chronic gastrointestinal disorders, or capsule swallowing difficulties, or prior surgical resection of intestinal segments;
14. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
RP2D | Up to 30 days after the first dose
  The RP2D is defined as the dose level chosen for phase II study, based on safety, tolerability, efficacy, collected during the dose escalation study of SHR0302.
Incidence and severity of AEs and SAEs | The first dose until 30 days after last dose
  To evaluate the safety and tolerability of SHR0302 in patients with PTCL in terms of AEs and SAEs as Assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided